CLINICAL TRIAL: NCT03398642
Title: Influence of Lifestyle Redesign® on Health, Social Participation, Leisure and Mobility of Older French-Canadians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Université de Montréal (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Research Centre on Aging, CIUSSS de l'Estrie-CHUS (Unknown); Université du Québec à Trois-Rivières (Other); University of Sheffield (Other)
Responsible Party: Principal Investigator, Mélanie Levasseur, Research Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-488; 126315 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2017-11-07; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Community-dwelling Older Adults
Keywords: Occupational therapy; Health promotion; Life Style; Quality of life; Aging; Aged; Community participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- French Lifestyle Redesign (Experimental): 16 older adults, 10 without and 6 with disabilities, participated to weekly 2-hour group sessions, including outings, and monthly 1-hour individual sessions led by a occupational therapist over 6-month period and promoting healthy lifestyle and involvement in meaningful activities.
  Interventions: Behavioral: French Lifestyle Redesign

INTERVENTIONS:
Behavioral: French Lifestyle Redesign — Lifestyle Redesign® is a preventive occupational therapy intervention designed to promote meaningful and healthy activities. The French-Canadian Lifestyle Redesign® intervention was led by an occupational therapist (OT) who took the University of Southern California 6-hour online introductory training course and was supervised on a weekly basis. Weekly 2-hour group sessions were held over a six-month period.These sessions were based on 12 modules (e.g. occupation, health and aging; transportation and occupation) from the 2nd edition of the Lifestyle Redesign® Manual and involved didactic presentations, peer exchanges, reflective exercises, direct experience and personal exploration. Every month, one group outing was targeted and individual meetings with the OT were planned.

SUMMARY:
To address population aging, health professionals, including occupational therapists, need to engage in effective interventions. The preventive occupational therapy intervention called Lifestyle Redesign® empowers older adults to regularly perform healthy and fulfilling activities. Lifestyle Redesign® has been shown to benefit physical and mental health and be cost-effective.

This pilot study explored the influence of Lifestyle Redesign® on older French- Canadians' health, social participation, leisure and mobility. Method: A mixed-method design was used with 16 participants (10 women) aged 65-90 (76.4±7.6 y), 10 without and 6 with disabilities. Health, social participation, leisure and mobility questionnaires were administered before and after the 6-month intervention, as well as 3 and 6 months post-intervention. Semi-directed interviews were also conducted.

DETAILED DESCRIPTION:
Study Design and Participants This pilot study used a mixed-method concurrent triangulation design including a pre-experimental component [pre-test (T1), post-test (T2) and follow-ups (T3 and T4)] and an exploratory descriptive qualitative clinical study with a sample of 16 community-dwelling older adults with and without disability. A sample size of 16 participants allowed detection of a standardized difference of 0.75 or greater between two means according to paired bilateral t tests based on a significance level of 5% and power of 80%. This difference was sufficient in a study that explored the influence of another intervention on leisure and life-space mobility. This sample size also allowed in-depth exploration and data saturation. Eligibility criteria were: 1) aged 65 and over, 2) no or mild (group 1) or moderate or severe (group 2) loss of autonomy, 3) normal cognitive functions, 4) living in a conventional or residential home for semi-independent seniors, and 5) French-speaking. Participants were recruited from a previous study of people attending a day hospital and day center in a Health and Social Services Centre (HSSC) in Quebec (Canada), and from people living in a residence. The Research Ethics Committee of the Eastern Townships HSSC approved the study (2015-488).

Data Collection Procedures Participants were recruited until the predetermined sample size (n=16+3, anticipating possible attrition) was reached. All participants signed an informed consent form and were met individually at home by a research assistant or occupational therapy student specially trained to administer the questionnaires. An experienced research assistant conducted the qualitative interviews. At T1, one sociodemographic and eight outcome questionnaires, four reported here and others elsewhere (Trépanier et al., in preparation), were administered in approximately 120 minutes. Following the six-month intervention period, participants answered the same outcome questionnaires (T2) and, about one month later, had a face-to-face semi-structured individual interview lasting about 90 minutes. All interviews were digitally audiotaped, transcribed and verified with respect to the wording used by participants. After the first few interviews, two authors (MB and ML) discussed and adjusted the questions for subsequent interviews. Finally, three (T3) and six (T4) months after the end of the intervention, participants answered the same questionnaires again.

Intervention In the present study, the French-Canadian Lifestyle Redesign® intervention was led by an occupational therapist (OT) who took the University of Southern California 6-hour online introductory training course. The OT was also supervised on a weekly basis by an academic OT specializing in health promotion and clinical research, and having a good knowledge of the intervention (highly involved in the translation). This supervision allowed the OT to have regular feedback on her role and intervention. Weekly 2-hour group sessions were held over a six-month period between August 2015 and March 2016. These sessions were based on 12 modules (e.g. occupation, health and aging; transportation and occupation) from the 2nd edition of the Lifestyle Redesign® Manual and involved didactic presentations, peer exchanges, reflective exercises, direct experience and personal exploration. Every month, one group outing was targeted and individual meetings with the OT were planned. These meetings aimed to help participants integrate the group session content and engage in personalized meaningful activities. In the group with participants having moderate or severe loss of autonomy, assistance to the OT was provided by one or two volunteers during respectively group sessions or outings.

Outcome Variables and Tools Data on health, social participation, leisure and life-space mobility were collected with four questionnaires. The 36-item Short Form Health Survey (SF-36) comprises 36 items covering eight domains related to physical and mental health. The SF-36 has good psychometric properties and is widely used in research, including previous Lifestyle Redesign® studies. The Social Participation Scale estimates the frequency of participation in 10 community activities and has shown good internal consistency. The Leisure Profile assesses involvement in leisure activities, attitudes toward leisure, and difficulties that might influence leisure activities; it has acceptable interrater and test-retest reliability. The Life-Space Assessment (LSA) measures life-space mobility and, more specifically, the range, independence, and frequency of movement over the preceding four weeks. The LSA presents good construct validity with observed physical performance and self-reported function and good sensitivity to change. Finally, a semi-structured interview guide validated by 5 qualitative research experts and pretested was used to explore the effect of Lifestyle Redesign®. Examples of questions were: 'Tell me about your experience with the program'; 'If applicable, how have your activities changed as a result of the program?' and 'How did the program help you make this change?' Data Analysis The participants' sociodemographic characteristics and outcomes were analyzed using descriptive statistics. Scores were compared with the Friedman test followed by the Wilcoxon signed rank test but for all participants and, in an exploratory manner, for participants of each group separately. Because of the exploratory nature of this study and the influence of seasonal variations on Quebecers' health, social participation, leisure and mobility, changes at any of the post-intervention measurement times with a p value < 0.05 were consider to be potentially attributable to the intervention. Interview transcripts underwent thematic content analysis using mix extraction grids. Themes that emerged from the interview content were organized and renamed according to the Human Development Model-Disability Creation Process, a model of human development and disability. The coauthor cocoded one-third of the data and closely supervised the analysis that underwent adjustement to reach a consensus. For parsimony with respect to the quantitative results, themes presented in this paper focus on health, social participation, leisure and mobility. Analyses were conducted using SPSS Statistics (v18) or NVivo (v10).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 and over
2. Normal cognitive functions
3. Living in a conventional or residential home for semi-independent seniors
4. French-speaking -

Exclusion Criteria:

1. Moderate or severe cognitive impairment [score < 17 Adult Lifestyles and Function Interview-Mini-Mental State Examination (ALFI-MMSE)]
2. Moderate or severe language impairment -

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
36-item Short Form Health Survey (SF-36) version 2, for the assessment of changes in physical and Mental Health from before at 6, 9 and 12 months after the intervention | Baseline, 6, 9, 12 months
  Full scale name: 36-item Short Form Health Survey (SF-36) version 2. Construct: The SF-36v2® assesses the health-related quality of life (HRQOL). Scale ranges: 0-100 for the scoring of eight health domains: (1-Physical Functioning, 2-Role Physical, 3-Bodily Pain, 4-General Health, 5-Vitality, 6-Social Functioning, 7-Role Emotional, 8-Mental Health) and of the Physical Component Summary (PCS) and Mental Component Summary (MCS), which can be calculated when seven scale scores are available and, for the PCS, when the Physical Functioning scale is not missing and for the MCS, when the Mental Health scale is not missing. A unique scoring algorithm is apply to the calculation of the summary scores depending upon which particular scale score is missing from the eight scale profiles. Higher score indicates better health.

SECONDARY OUTCOMES:
Social Participation Scale, for the assessment of change in the frequency of participation in ten community activities from before at 6, 9 and 12 months after the intervention | Baseline, 6, 9, 12 months
  Full scale name (in French): "Fréquence de réalisation de 10 activités sociales et communautaires". Construct: This questionnaire includes questions (n = 10) to assess the frequency of participation in 10 (social or leisure) activities in the past year. Scale ranges: 0-200. Calculation of the total score: The values obtained in the 10 questions are summed, which are: almost every day = 20, at least once a week = 6, at least once a month = 2, less than once a month = 1, never = 0. Higher score indicates a greater frequency of participation.
Leisure Profile, for the assessment of change in leisure, attitudes and limitations from before at 6, 9, and 12 months after the intervention | Baseline, 6, 9, 12 months
  Full scale name: Leisure Profile (in French: "Profil du loisir"). Construct: This tool assesses leisure, residual capacities and limitations. Items evaluated in connection to involvement in leisure activities: 1-Level of interest,2- Frequency of practice, 3-Desire to modify the practice and 4-Frequency. The maximum score determined for each item is 30, except for the desire to modify the practice the maximum score is 15. Items evaluated in connection to attitudes: 1-positive, 2-negative. The maximum total score with subscales summed is 34 (subscale scores for each item: 17). Items evaluated in connection to difficulties: 1-Impairments, 2- Influence on leisure (maximum score for each: 17), 3- Physical environment obstacles, 4- Influence on leisure (maximum score for each: 5), 5-Social environment obstacles, 6- Influence on leisure (maximum score for each: 6). Higher score indicates greater involvement in leisure activities, positive attitude toward leisure, or fewer difficulties.
French-Canadian version of Life-Space Assessment, for the assessment of change in range, independence and frequency of movement in the 4 last weeks from before at 6, 9 and 12 months after the intervention | Baseline, 6, 9, 12 months
  Full scale name: French-Canadian version of Life-Space assessment (LSA-F). Construct: The LSA assesses the range, independence, and frequency of movement over the 4 weeks. The LS-maximum score is the maximum mobility area reached by the person with or without technical or human assistance. The LS-Assisted score is the maximum mobility area reached by the person with technical assistance only. The LS-Independent score is the maximum mobility area reached by the person without technical and human assistance. For these three measures, the maximum score is 5. For each area, the area level is multiplied by the frequency and level of independence. The LS-C composite score is the sum of the result obtained for each of the 5 mobility areas. Higher score indicate better range, independence and frequency of movement over the last 4 weeks.
Exploration of the influence of the French Lifestyle Redesign | About one month after the intervention
  After the experimentation: Qualitative interviews with all of the participants to explore the influence of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Levasseur, Principal Investigator — Université de Sherbrooke, Centre de recherche sur le vieillissement

IPD SHARING:
Plan to Share IPD: Undecided